CLINICAL TRIAL: NCT02783287
Title: The Impact of Text Messaging on Medication Adherence and Exercise Regimen Among Post-myocardial Infarction Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Waterloo (Other)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Associate Professor of Medicine at Harvard Medical School, Associate Physician in the Division of Pharmacoepidemiology and Pharmacoeconomics and the Hospitalist Program at Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20980
Record Dates: First submitted 2016-01-07; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Myocardial Infarction
Keywords: Exercise adherence; Medication adherence; Mobile health; Cardiac rehabilitation
MeSH Terms: conditions — Myocardial Infarction; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Medication text message (Experimental): Once daily text message reminder.
  Interventions: Behavioral: Text message reminder for medication adherence
- Exercise text message (Experimental): 4x daily text message reminder.
  Interventions: Behavioral: Text message reminder for exercise regimen
- Usual care, medication adherence (No Intervention): Usual care for medication adherence.
- Usual care, exercise regimen (No Intervention): Usual care for exercise regimen.

INTERVENTIONS:
Behavioral: Text message reminder for medication adherence — Patients randomized to this arm receive one text message per day (at the scheduled time) reminding them to take their medication.
  Arms: Medication text message
Behavioral: Text message reminder for exercise regimen — Patients randomized to this arm receive 4 daily text messages reminding them to exercise for 30 minutes per day.
  Arms: Exercise text message

SUMMARY:
The purpose of this study is to assess the impact of text message reminders on adherence to medications and exercise in patients recently discharged from the hospital after a myocardial infarction (MI).

DETAILED DESCRIPTION:
The Impact of Text Messaging on Medication Adherence and Exercise Regimen among Post-Myocardial Infarction Patients includes two single-center randomized control trials to assess the impact of text message reminds on adherence to medications and exercise regimen in patients recently discharged from the hospital after MI.

Recruitment conducted at Cambridge Cardiac Rehabilitation in Ontario, Canada for both the medication adherence and exercise trial. Potential study subjects are evaluated for inclusion and exclusion criteria, give written informed consent, and are randomized, in a 1:1 ratio, to either intervention or usual care (control).

Patients randomized to the intervention arm in the medication adherence trial receive an automated text message once per day at the time they are prescribed to take their medication. The text message does not contain any personal or pharmacological information.

Patients randomized to the intervention arm in the exercise adherence trial receive four text messages per day at 7:30 am, 12:00 pm, 6:00 pm, and 9:00 pm, reminding them to exercise for 30 minutes per day as per their health care provider.

ELIGIBILITY:
Inclusion Criteria:

* Post-MI hospital discharge within 2 weeks
* Enrolled in cardiac rehabilitation
* Prescribed anti-platelets, beta-blockers, ACE-inhibitors or ARBs, and/or statins on 1x/day regimen (for medication adherence trial)
* Prescribed exercise regimen (for exercise trial)
* Ability to read and write English
* Possession of a cell phone with text messaging capability

Exclusion Criteria:

* Age < 18
* Incarcerated individuals
* Unable to read and write English
* Not in possession of a cell phone
* Patients prescribed medication regimen > 1x/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 12 months
  Average medication adherence over 12 months after randomization, assessed with self-reported logs
Exercise frequency | 12 months
  Average frequency of exercise over 12 months after randomization, assessed with self-reported logs

SECONDARY OUTCOMES:
Exercise duration | 12 months
  Average duration of exercise assessed by BRUCE protocol
Full medication adherence | 12 months
  Average medication adherence over 12 months greater than .80

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Center for Healthcare Delivery Sciences, Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pandey A, Krumme AA, Patel T, Choudhry NK. The Impact of Text Messaging on Medication Adherence and Exercise Among Postmyocardial Infarction Patients: Randomized Controlled Pilot Trial. JMIR Mhealth Uhealth. 2017 Aug 3;5(8):e110. doi: 10.2196/mhealth.7144. PMID 28778843